CLINICAL TRIAL: NCT03909009
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Pain, Fatigue, Quality of Life, Cognitive Function and Mood in Fibromyalgia
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, İbrahim Bilir, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14032019
Record Dates: First submitted 2019-03-17; First posted 2019-04-09 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, neuronavigated-rTMS, pain, stiffness, fatigue
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Transcranial Magnetic Stimulation; Neuronavigation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS (Active Comparator): Group 1 will receive high frequency repetitive transcranial magnetic stimulation (10hz-HF-rTMS) A total 14 sessions of HF-rTMS, 10 sessions daily (5 days/week, 2 weeks) and 4 sessions weekly (1 day/week, 4 weeks).
  Interventions: Device: rTMS + Neuronavigation
- Sham rTMS (Sham Comparator): Group 2 will receive sham stimulation. A total 14 sessions of sham-rTMS, 10 sessions daily (5 days/week, 2 weeks) and 4 sessions weekly (1 day/week, 4 weeks).
  Interventions: Device: rTMS + Neuronavigation

INTERVENTIONS:
Device: rTMS + Neuronavigation — Repetitive Transcranial Magnetic Stimulation (Neuro-MS/D) + Neural Navigator

SUMMARY:
This study aims to evaluate the effectiveness of 10 Hz neuronavigated repetitive transcranial magnetic stimulation (rTMS) to the left dorsolateral prefrontal cortex (DLPFC) on pain, stiffness, fatigue, depression/anxiety, quality of life and cognitive functions in fibromyalgia syndrome (FMS).

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, double-blind, sham-controlled study in two-arm parallel-group design. Twenty participants will be randomized into 2 groups. Randomization will be performed using computer-generated block randomization with 1:1 allocation between the active rTMS group (Group 1) and the sham-control group (Group 2). Group 1 will receive high frequency repetitive transcranial magnetic stimulation (10hz-HF-rTMS)-A total 14 sessions of HF-rTMS, 10 sessions daily (5 days/week, 2 weeks) and 4 sessions weekly (1 day/week, 4 weeks). Group 2 will receive sham stimulation-A total 14 sessions of sham-rTMS, 10 sessions daily (5 days/week, 2 weeks) and 4 sessions weekly (1 day/week, 4 weeks).All patients will be evaluated with pain severity (VAS-10mm),stiffness severity (VAS-10mm), Fibromyalgia Impact Questionnaire (FIQ), Fatigue Severity Scale (FSS), Hospital Depression Anxiety Scale (HADS), Addenbrook Cognitive Examination-revised version (ACE-R).Patients will be questioned for the safety of treatment. Available drug therapies will be continued in both groups. Patients and clinical raters will be blinded to treatment. All patients will be reviewed by the investigator in terms of rTMS treatment safety and motor threshold determination before each treatment session and observed for possible side effects after treatment. All side effects will be recorded. Magnetic stimulation will be applied using Neurosoft-Neuro MS/D with a figure-of-eight-shaped coil. rTMS therapy will be applied under the guide of neuronavigation with the following parameters: target-left DLPFC, with the %90 of the RMT, 10 Hz stimulation for 5 seconds intervals (on) with 25 seconds inter-train intervals (off), 15 minutes, 1500 pulses.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age between 18-65 years)
* Diagnosis of fibromyalgia syndrome according to 2016 Fibromyalgia diagnostic criteria
* The mean pain intensity is VAS ≥ 4/10
* Stable treatment for at least last 3 months
* Patients accepting participation by signing an informed consent form

Exclusion Criteria:

* To have a clinical condition to be contraindicated for TMS (metallic implant, cardiac pace, pregnancy, lactation, epilepsy, head trauma, history of cranial operation...)
* The presence of malignancy
* Systemic rheumatic diseases
* Major orthopedic / neurological problems that limit daily life activities
* Alcohol or drug addiction
* Major depression / personality disorder history
* Have received TMS treatment before
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Aşkın, Assoc. Prof., Study Director — Izmir Katip Çelebi University Faculty of Medicine
Locations (1):
- Izmir Katip Çelebi University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Klein MM, Treister R, Raij T, Pascual-Leone A, Park L, Nurmikko T, Lenz F, Lefaucheur JP, Lang M, Hallett M, Fox M, Cudkowicz M, Costello A, Carr DB, Ayache SS, Oaklander AL. Transcranial magnetic stimulation of the brain: guidelines for pain treatment research. Pain. 2015 Sep;156(9):1601-1614. doi: 10.1097/j.pain.0000000000000210. PMID 25919472
- [Background] Knijnik LM, Dussan-Sarria JA, Rozisky JR, Torres IL, Brunoni AR, Fregni F, Caumo W. Repetitive Transcranial Magnetic Stimulation for Fibromyalgia: Systematic Review and Meta-Analysis. Pain Pract. 2016 Mar;16(3):294-304. doi: 10.1111/papr.12276. Epub 2015 Jan 12. PMID 25581213
- [Background] Hou WH, Wang TY, Kang JH. The effects of add-on non-invasive brain stimulation in fibromyalgia: a meta-analysis and meta-regression of randomized controlled trials. Rheumatology (Oxford). 2016 Aug;55(8):1507-17. doi: 10.1093/rheumatology/kew205. Epub 2016 May 5. PMID 27150193
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Saltychev M, Laimi K. Effectiveness of repetitive transcranial magnetic stimulation in patients with fibromyalgia: a meta-analysis. Int J Rehabil Res. 2017 Mar;40(1):11-18. doi: 10.1097/MRR.0000000000000207. PMID 27977465
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Baudic S, Attal N, Mhalla A, Ciampi de Andrade D, Perrot S, Bouhassira D. Unilateral repetitive transcranial magnetic stimulation of the motor cortex does not affect cognition in patients with fibromyalgia. J Psychiatr Res. 2013 Jan;47(1):72-7. doi: 10.1016/j.jpsychires.2012.09.003. Epub 2012 Oct 15. PMID 23079535
- [Background] Tekin A, Özdil E, Güleken MD, İlişer R, Bakım B, Öncü J, et al. Efficacy of HighFrequency [10 Hz] Repetitive Transcranial Magnetic Stimulation of the PrimaryMotor Cortex in Patients with Fibromyalgia Syndrome: A Randomized, DoubleBlind, Sham-Controlled Trial. Journal of Musculoskeletal Pain. 2014;22(1):20-26.
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Derived] Bilir I, Askin A, Sengul I, Tosun A. Effects of High-Frequency Neuronavigated Repetitive Transcranial Magnetic Stimulation in Fibromyalgia Syndrome: A Double-Blinded, Randomized Controlled Study. Am J Phys Med Rehabil. 2021 Feb 1;100(2):138-146. doi: 10.1097/PHM.0000000000001536. PMID 32701637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Physical Medicine and Rehabilitation (PMR) outpatient clinics of a university hospital.
Pre-assignment Details: Twenty-eight patients were evaluated for participation in the study. Eight patients were excluded.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.70 (9.06) | 43.80 (9.37) | 45.25 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 10 | 10 | 20
Visual Analog Scale-Pain [Mean (Standard Deviation); unit: units on a scale] — The severity of the pain at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no pain, 10=severe pain)
  units on a scale | 7.20 (1.75) | 7.40 (1.35) | 7.30 (1.52)
Visual Analog Scale-Stiffness [Mean (Standard Deviation); unit: units on a scale] — The severity of the stiffness at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no stiffness, 10=severe stiffness)
  units on a scale | 7.40 (1.58) | 7.60 (1.17) | 7.50 (1.35)
Fibromyalgia Impact Questionnaire [Mean (Standard Deviation); unit: scores on a scale] — Functional health status and quality of life of the participants were assessed with the Fibromyalgia impact questionnaire, which measures 10 different features (physical functioning, missed days of work, depression, anxiety, feeling good, morning tiredness, pain, stiffness, fatigue, and well-being over the past week). The total Fibromyalgia impact questionnaire score is maximum 80 points. Higher scores indicate lower functionality level.
  scores on a scale | 65.86 (8.27) | 66.44 (11.40) | 66.15 (9.69)
Fatigue Severity Scale [Mean (Standard Deviation); unit: scores on a scale] — Severity of fatigue was evaluated with Fatigue severity scale, a 9-item self-report questionnaire scale. Each item of this scale consists of statements that are scored on a seven-point Likert type scale ranging from 1 to 7. Total Fatigue severity scale score is calculated as the mean value of nine items. Higher scores indicate higher fatigue severity. (Total score range: 1-7)
  scores on a scale | 5.28 (1.23) | 6.08 (1.11) | 5.68 (1.20)
Hospital Anxiety and Depression Scale [Mean (Standard Deviation); unit: scores on a scale] — HADS is an assessment tool developed to identify the risk of anxiety and depression and measure its level and change of severity. Its subscales are anxiety and depression. It contains 14 questions in total, including 7 (odd numbers) measuring anxiety and 7 (even numbers) measuring depression. The lowest and highest total score that a person can obtain from this scale are 0 and 42, respectively. High scores are associated with a worse psychiatric condition.
  scores on a scale | 19.30 (8.14) | 22.90 (5.61) | 21.10 (7.04)
Addenbrook Cognitive Examination Revised [Mean (Standard Deviation); unit: scores on a scale] — Addenbrook Cognitive Examination Revised (ACE-R): ACE-R is a brief cognitive test that consists of 5 basic sections: attention and orientation, memory, verbal fluency, language and visual-spatial abilities. Total score that can be obtained is 0-100. Higher scores are associated with a better cognitive state.
  scores on a scale | 62.50 (18.80) | 76.90 (11.17) | 69.70 (16.76)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale-Pain
Description: The severity of the pain at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no pain, 10=severe pain) Higher scores mean a worse outcome.
Time Frame: in the second week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
units on a scale | 5.30 (2.11) | 6.80 (1.69)

2. Secondary Outcome: Visual Analog Scale-Pain
Description: as for outcome 1
Time Frame: in the sixth week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
units on a scale | 5.70 (2.63) | 6.70 (1.83)

3. Secondary Outcome: Fibromyalgia Impact Questionnaire
Description: Functional health status and quality of life of the participants were assessed with the Fibromyalgia impact questionnaire, which measures 10 different features (physical functioning, missed days of work, depression, anxiety, feeling good, morning tiredness, pain, stiffness, fatigue, and well-being over the past week). The total Fibromyalgia impact questionnaire score is maximum 80 points. Higher scores indicate lower functionality level.
Time Frame: in the sixth week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
score on a scale | 51.71 (22.17) | 56.02 (22.57)

4. Other Pre Specified Outcome: Visual Analog Scale-Stiffness
Description: The severity of the stiffness at rest was assessed on a 10 cm visual analog scale (Total score: 0-10)(0=no stiffness, 10=severe stiffness) Higher scores mean a worse outcome.
Time Frame: in the second week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
units on a scale | 5.10 (2.13) | 6.60 (1.96)

5. Other Pre Specified Outcome: Fibromyalgia Impact Questionnaire
Description: as for outcome 3
Time Frame: in the second week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
score on a scale | 48.35 (16.64) | 54.39 (15.47)

6. Other Pre Specified Outcome: Fatigue Severity Scale
Description: Severity of fatigue was evaluated with Fatigue severity scale, a 9-item self-report questionnaire scale. Each item of this scale consists of statements that are scored on a seven-point Likert type scale ranging from 1 to 7. Total Fatigue severity scale score is calculated as the mean value of nine items. Higher scores indicate higher fatigue severity. (Total score range: 1-7)
Time Frame: in the sixth week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
score on a scale | 4.89 (1.59) | 5.39 (1.62)

7. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale
Description: Hospital anxiety and depression scale is an assessment tool developed to identify the risk of anxiety and depression and measure its level and change of severity. Its subscales are anxiety and depression. It contains 14 questions in total, including 7 (odd numbers) measuring anxiety and 7 (even numbers) measuring depression. The lowest and highest total score that a person can obtain from this scale are 0 and 42, respectively. High scores are associated with a worse psychiatric condition.
Time Frame: in the sixth week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
score on a scale | 18.80 (7.82) | 17.60 (10.68)

8. Other Pre Specified Outcome: Addenbrook Cognitive Examination Revised
Description: Addenbrook Cognitive Examination-Revised is a brief cognitive test that consists of 5 basic sections: attention and orientation, memory, verbal fluency, language and visual-spatial abilities. Total score that can be obtained is 0-100. Higher scores are associated with a better cognitive state.
Time Frame: in the sixth week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
score on a scale | 66.50 (19.67) | 81.40 (7.79)

ADVERSE EVENTS:
Time Frame: 6 weeks (Between the start of the study and the day when the last outcome measure is evaluated)
Groups:
- Active rTMS: Group 1 will receive HF rTMS treatment daily from Monday to Friday in first 2 weeks. After first 2 weeks there will be sessions once a week for 1 month.
  There will be 14 sessions in total.
  rTMS + Neuronavigation: Repetitive Transcranial Magnetic Stimulation (Neuro-MS/D) + Neural Navigator
- Sham rTMS: Group 2 will receive sham daily from Monday to Friday in first 2 weeks. After first 2 weeks there will be sessions once a week for 1 month.
  There will be 14 sham sessions in total.
  rTMS + Neuronavigation: Repetitive Transcranial Magnetic Stimulation (Neuro-MS/D) + Neural Navigator
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Current study has several limitations: First is the relatively small sample size. Second, we didn't use sham stimulation probe. Third, our patients only consisted of female gender.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT03909009/Prot_SAP_000.pdf